CLINICAL TRIAL: NCT04880889
Title: Study Phase III, Randomized, Double-dummy, Placebo Controlled, Single-center, of Regarding the Non-inferiority of the Medication BL3000, When Compared to Pantogar® Treatment of Telogen Effluvium in Women.
Brief Title: BL3000 Compared to Pantogar® in the Treatment of Telogen Effluvium in Women.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP165762
Record Dates: First submitted 2021-03-01; First posted 2021-05-11 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Telogen Effluvium
Keywords: loss of hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Study phase III, randomized, double-dummy, placebo controlled, single-center, of regarding the non-inferiority of the medication BL3000, when compared to Pantogar® treatment of telogen effluvium in women.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL 3000 (active) and Pantogar matching Placebo (Experimental): One capsule, once a day for 180 days for BL3000 and one capsule three times a day for Pantogar-Placebo.
  Interventions: Drug: BL 3000; Drug: Pantogar - Placebo
- Pantogar and BL3000 matching placebo (Active Comparator): One capsule, three times a day for 180 days
  Interventions: Drug: Reference Pantogar; Drug: BL3000 Placebo

INTERVENTIONS:
Drug: BL 3000 — capsule 500 mg
  Arms: BL 3000 (active) and Pantogar matching Placebo
Drug: Reference Pantogar — capsule
  Arms: Pantogar and BL3000 matching placebo
Drug: BL3000 Placebo — capsule 500 mg
  Arms: Pantogar and BL3000 matching placebo
Drug: Pantogar - Placebo — capsule
  Arms: BL 3000 (active) and Pantogar matching Placebo

SUMMARY:
Study phase III, randomized, double-dummy, placebo controlled, single-center, of regarding the non-inferiority of the medication BL3000, when compared to Pantogar® treatment of telogen effluvium in women.

Research product: BL3000. Reference product: Pantogar® List of Study Center: MAIN INVESTIGATOR STUDY CENTER FONE Medcin Skin Institute Sérgio Schalka 11 36835357

DETAILED DESCRIPTION:
Study phase III, randomized, double-dummy, placebo controlled, single-center, of regarding the non-inferiority of the medication BL3000, when compared to Pantogar® treatment of telogen effluvium in women. 326 female patients will be recruited for the study. They will be aged from 18 to 45 years old, not menopausal, diagnosed with telogen effluvium proven by Trichoscan, who meet the inclusion criteria and do not meet the exclusion criteria and who sign the Informed Consent Form.

Patients will be divided into two treatment groups according to randomization:

Group I: 163 patients will receive treatment with the medication BL3000 and matching placebo of pantogar.

Group II: 163 patients will receive treatment with the reference drug (Pantogar®) and matching placebo of BL3000.

The patients will participate in the study for a period of 199 (one hundred and ninety-nine) days, using of the investigational or comparative product for 180 (one hundred and eighty) days,

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged from 18 to 45 years old;
2. Clinical/trichological evidence of telogen effluvium, assessed using the Telogen Index. 3. Participants will be eligible if they have a rate strand of hair ≥ 20% of the total quantified by Thrichoscan measurement in the central-parietal region;
3. Complaint of hair loss for at least 3 months prior to screening;
4. Agreement to obey the procedures and requirements of the protocol and to attend the Research Institution on the day (s) and time (s) determined for the evaluations;
5. Signature of the Informed Consent Form; SAW. Agreement to use an acceptable non-hormonal contraceptive method throughout the period of treatment and up to 60 days after the end of the study;
6. Serum creatinine within the normal range;
7. Relationship between AST / ALT transaminases ≤ 2.5x the upper limit of normal

Exclusion Criteria:

1. Pregnancy or pregnancy risk;
2. Lactation;
3. Childbirth occurred in the last 12 months;
4. Patient who has undergone surgical procedures or has suffered trauma in the last 6 months;
5. History of bleeding events in the last 6 months, SAW. Clinical evidence of female androgenic alopecia or alopecia areata;
6. Patients with signs of menopause: menstrual irregularities or cycle failure, signs of climacteric;
7. Laboratory evidence of thyroid diseases (variation in TSH and / or free T4 values outside normal limits);
8. Clinical evidence of ovarian or adrenal endocrine disorders (polycystic ovaries, hirsutism, menstrual irregularities);
9. History or presence of systemic autoimmune disease;
10. Start or end of hormone therapy within 6 months before randomization;
11. Deficiency diseases;
12. Introduction, change or interruption of a hormonal contraceptive method in the last 6 months before randomization;
13. Introduction of a restrictive diet in the last 03 months before randomization;
14. Use of any continuous medication;
15. Diabetes, chronic consuming disease, malabsorptive syndrome or diseases of the gastrointestinal tract;
16. Infectious or chronic fever;
17. Psychiatric/psychological illnesses, such as depression, anxiety or obsessive disorders;
18. Clinical and / or laboratory evidence of anemia or ferropenia; (Hb <12 g / dL and Ferritin <40 g / L);
19. Hair treatment to control hair loss (including shampoo, conditioner, lotions);
20. Hair growth agent treatment within 3 months before randomization;
21. Concomitant use of drugs that cause hair loss;
22. Patient with a history of allergic reaction or hypersensitivity to any formulation ingredients;
23. Other conditions considered by the evaluating physician to be reasonable for disqualifying the participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate difference of anagen hairs at 180 days (FA vf [%]) from baseline rate (FA vi [%]), in participants of each treatment group. | 180 days
  Assess the non-inferiority of the effectiveness of the BL3000 drug compared to the drug.
  The counting of anagen and telogen performed by phototrichogram in the initial and final experimental times, with the calculation proposed according to the protocol below:
  The primary variable of efficacy will be the rate of anagen hairs (FA) (%), 45.90 and 180 days in relation to the beginning, between the two arms of treatment (test versus control). Calculated as follows:
  FA (vi): result of anagen (%) on visit 04 (T0); FA (vf): result of anagen (%) on visit 10 (T182). Response rate of anagen (%), FA = (FA (vf)-FA (vi)).

SECONDARY OUTCOMES:
Difference of the total count of strand hair per mm² (density) at the experimental time frames, compared to the baseline evaluation, in participants of each treatment group. | 45,90 and 180 days
  Difference of the density of the strand hair, in a given area (units per mm2), measured by phototrichogram in the experimental times, compared to the baseline measurement
Difference of the number of anagen hairs per mm² (density) at the experimental time frames, compared to the baseline evaluation, in participants of each treatment group. | 45,90 and 180 days
  Difference of the density of anagen hairs, in a given area (units per mm2), measured by phototrichogram in the experimental times, compared to the baseline measurement
Difference of the number of telogen hairs per mm² (density) at the experimental time frames, compared to the baseline evaluation, in participants of each treatment group. | 45,90 and 180 days
  Difference of the density of telogen hairs, in a given area (units per mm2), measured by phototrichogram in the experimental times, compared to the baseline measurement
Difference of the anagen/telogen hair ratio at the experimental times frames, compared to the baseline evaluation, in participants of each treatment group. | 45,90 and 180 days
  Difference of the anagen/telogen hair ratio, in a given area (units per mm2), measured by phototrichogram in the experimental times, compared to the baseline measurement
Difference of the strand hair thickness (mm²) at the experimental time frames, compared to the baseline evaluation, in participants of each treatment group. | 45,90 and 180 days
  Difference of the thickness of strand hairs, measured by phototrichogram in the experimental times, compared to the baseline measurement
Proportion of "Excellent" and "Very good" change of the telogen effluvium, as assessed by the investigator, comparing photographs taken at final visit and baseline visit, in participants of each treatment group. | 180 days
  Analysis photographs taken during the initial and final visits, the opinion of the evaluator, regarding the improvement of the telogen effluvium:
  1. - Excellent;
  2. - Very good;
  3. - Good;
  4. - Regular
  5. - Bad. Analysis global assessment of the investigator, the X2 test will be used to make comparisons between groups. The proportion of Excellent and Very good for Researcher question will be analyzed, the confidence interval with 95% confidence for p1 - p2 will be constructed from the sample distribution of the sample proportion, where p2 is the proportion of Excellent and Very good by Pantogar for Researcher question and p1 is that of the test drug.
Proportion of "Much better" and "best" change, based on the participant's subjective assessment, from each treatment group, using a Likert scale. | 45,90 and 180 days
  Participants will present their opinion on the effectiveness of the treatment, using a Likert scale from 1 to 4:
  Considering the evolution of the treatment, what is your opinion about the amount of hair strands at the end of the treatment.
  1 - Much better; 2 - Best; 3 - No change and 4 - Worse. To analyze Subjective evaluation of the patient, the X2 test will be used to make comparisons between groups.
  The proportion of Much better and Best for patient question will be analyzed, the confidence interval with 95% confidence for p1 - p2 will be constructed from the sample distribution of the sample proportion, where p2 is the proportion of Very best and Best of Pantogar for patient question and p1 is that of the test drug.
Number of participants with treatment-related adverse events in each treatment group | 180 days
  Safety and tolerability evaluation based on the occurrence of adverse events in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Schalka, Principal Investigator — Medcin Instituto da Pele